CLINICAL TRIAL: NCT02734550
Title: (1,3)-β-D-glucan Based Diagnosis of Invasive Candida Infection Versus Culture Based Diagnosis in Patients With Severe Sepsis or Septic Shock
Brief Title: (1,3)-β-D-glucan Based Diagnosis of Invasive Candida Infection in Sepsis
Acronym: CandiSep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Sepsis Control and Care, Germany (Other)
Collaborators: Center for Clinical Studies, University Hospital Jena, Germany (Unknown); Dept. of Microbiology, University Hospital Erlangen, Germany (Unknown); Institute of Medical Statistics, Computer Sciences and Documentation, University Hospital Jena, Germany (Unknown); Federal Ministry of Education and Research, Berlin, Germany (Unknown); Associates of Cape Cod, Inc., East Falmouth, MA, USA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ZKSJ0087; 01EO1502 (Other Grant/Funding Number: Federal Ministry of Education and Research of Germany); U1111-1181-8724 (Registry Identifier: Universal Trial Number); DRKS00010285 (Registry Identifier: German Clinical Trial Register)
Record Dates: First submitted 2016-04-06; First posted 2016-04-12 (Estimated); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Severe Sepsis; Septic Shock
Keywords: Sepsis; Invasive Candida Infection; Biomarker; (1,3)-β-D-glucan; Antifungal therapy; Intensive care medicine; Critically ill
MeSH Terms: conditions — Sepsis; Shock, Septic; Critical Illness | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: investigator-initiated prospective, multicenter, randomized, open, and parallel group study
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Diagnosis of invasive candida infection according to standard of care.
  Interventions: Other: Standard of care
- (1,3)-β-D-glucan guidance (Experimental): Treatment according to BDG-result
  Interventions: Other: Standard of care; Other: (1,3)-β-D-glucan guided therapy

INTERVENTIONS:
Other: Standard of care — Patients are treated according to the ESCMID guidelines. Antifungal therapy is started if fungi are detected in the blood culture or other primary sterile body fluids.
Other: (1,3)-β-D-glucan guided therapy — Serum for (1,3)-β-D-glucan measurement is obtained after enrollment and 24 hours later. Antifungal therapy is started if at least one sample is 80 pg/ml or higher. If concomitantly taken microbiological cultures remain negative, antifungal therapy is continued only, if both (1,3)-β-D-glucan were at least 80 pg/ml. Blood cultures or other samples from primary sterile body fluids positive for fungi are treated with antifungals irrespective the (1,3)-β-D-glucan results.
  Arms: (1,3)-β-D-glucan guidance

SUMMARY:
This prospective randomized multicenter study evaluates whether the decision to prescribe antifungals guided by (1,3)-β-D-glucan in comparison to standard of care shortens time to antifungal therapy and reduces mortality in patients with severe sepsis or septic shock and a high risk of invasive candida infection.

DETAILED DESCRIPTION:
(1,3)-β-D-glucan is a component of the cell wall of many fungi including candida spp. and is present in the blood of patients with invasive candida infection (ICI). Several studies showed a good diagnostic accuracy (1,3)-β-D-glucan in predicting ICI. However, others have challenged (1,3)-β-D-glucan as a diagnostic tool in critically ill patients as many substances used in the intensive care unit might affect the results of the assay. The goal of this study is to investigate whether (1,3)-β-D-glucan can early identify sepsis patients in need of antifungal therapy. Patients randomized to the standard of care group receive antifungals depending on microbiological results according to current guidelines. Patients randomized to the BDG group receive antifungals depending on the (1,3)-β-D-glucan plasma concentration on day 1 and day after diagnosing sepsis. Therapy may be modified according to microbiological results.

ELIGIBILITY:
Inclusion Criteria:

* Severe sepsis or septic shock
* Onset of sepsis no longer than 24 hours
* Increased risk of invasive candida infection with at least one of the following criteria:

  * total parenteral nutrition ≥48 hours
  * abdominal surgery within the last 7 days
  * antimicrobial therapy for at least 48 hours within the last 7 days
  * Acute or chronic renal failure with renal replacement therapy
* Age ≥18 years
* Informed consent of the patient or legal representative or delayed consent process is started if patient is incapable of giving informed consent and no legal representative is available.

Exclusion Criteria:

* Pregnant or lactating women
* Ongoing invasive candida infection
* systemic antifungal therapy
* liver cirrhosis Child C
* cardiopulmonary bypass within the last 4 weeks
* treatment with immunoglobulins within the last 14 days
* immunosuppression (solid organ transplantation, AISA, leukopenia)
* participation in another intervention study
* no commitment to full therapy (i.e. DNR order)
* Infauste Prognose aufgrund von Nebenerkrankungen
* kin to or colleague of study personnel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
28 day mortality | 28 days

SECONDARY OUTCOMES:
28 day antifungal-free survival | 28 days
Candida Colonization | 14 days
  Candida colonization assessed by Candida Colonization Index
Time to antifungal therapy | 14 days
Duration of organ support | 14 days
Mean total SOFA score | 14 days
  Measure of organ dysfunction
ICU and hospital length of stay | Hospital length of stay
ICU and hospital mortality | Hospital length of stay
Adverse events | 14 days
Diagnostic performance of (1,3)-β-D-glucan in comparison to PCR and other experimental diagnostics | 2 days
Pharmacoeconomics | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Frank Bloos, MD, Ph.D., Principal Investigator — Jena University Hospital
Locations (18):
- Germany (18):
  - Hospital Augsburg, Augsburg
  - HELIOS Klinikum Bad Saarow, Bad Saarow
  - University Hospital Bonn, Bonn
  - Hospital Emden, Emden
  - University Hospital Erlangen, Erlangen
  - University Hospital Frankfurt, Frankfurt
  - University Hospital Göttingen, Göttingen
  - University Hospital Greifswald, Greifswald
  - University Hospital Halle, Halle
  - University Hospital Hamburg-Eppendorf, Hamburg
  - University Hospital Heidelberg, Heidelberg
  - Jena University Hospital, Jena
  - University Hospital Schleswig-Holstein, Kiel
  - University Hospital Leipzig, Leipzig
  - University Hospital Münster, Münster
  - Hospital Oldenburg, Oldenburg
  - Diakonie Klinikum, Siegen
  - University Hospital Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bloos F, Held J, Schlattmann P, Brillinger N, Kurzai O, Cornely OA, Thomas-Ruddel D. (1,3)-beta-D-glucan-based diagnosis of invasive Candida infection versus culture-based diagnosis in patients with sepsis and with an increased risk of invasive Candida infection (CandiSep): study protocol for a randomized controlled trial. Trials. 2018 Sep 4;19(1):472. doi: 10.1186/s13063-018-2868-0. PMID 30180873
- [Result] Bloos F, Held J, Kluge S, Simon P, Kogelmann K, de Heer G, Kuhn SO, Jarczak D, Motsch J, Hempel G, Weiler N, Weyland A, Druner M, Grundling M, Meybohm P, Richter D, Jaschinski U, Moerer O, Gunther U, Schadler D, Weiss R, Putensen C, Castellanos I, Kurzai O, Schlattmann P, Cornely OA, Bauer M, Thomas-Ruddel D; SepNet Study Group. (1 --> 3)-beta-D-Glucan-guided antifungal therapy in adults with sepsis: the CandiSep randomized clinical trial. Intensive Care Med. 2022 Jul;48(7):865-875. doi: 10.1007/s00134-022-06733-x. Epub 2022 Jun 16. PMID 35708758